CLINICAL TRIAL: NCT05119153
Title: Effects of Coffee Roasting on Blood Sugar Levels in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Gabriel Keith Harris, Associate Professor of Food Science, North Carolina State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16857
Record Dates: First submitted 2021-10-31; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Hyperglycemia
Keywords: coffee; glucose challenge; blood glucose levels
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, partial block, crossover design
Who Masked: Participant
Masking Description: Subjects provided placebo and coffee beverages in a color coded bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Comparator (Placebo Comparator): Placebo composed of water and caramel color.
  Interventions: Dietary Supplement: Placebo Comparator
- Light Roasted Coffee (Experimental): 12 oz light roast coffee beverage prepared at 55 g ground coffee/L water
  Interventions: Dietary Supplement: Light Roasted Coffee
- Medium Roasted Coffee (Experimental): 12 oz medium roast coffee beverage prepared at 55 g ground coffee/L water
  Interventions: Dietary Supplement: Medium Roasted Coffee
- Dark Roasted Coffee (Experimental): 12 oz dark roast coffee beverage prepared at 55 g ground coffee/L water
  Interventions: Dietary Supplement: Dark Roasted Coffee

INTERVENTIONS:
Dietary Supplement: Placebo Comparator — Placebo designed to mimic coffee color.
  Arms: Placebo Comparator
Dietary Supplement: Light Roasted Coffee — 12 oz light roast coffee
  Arms: Light Roasted Coffee
Dietary Supplement: Medium Roasted Coffee — 12 oz medium roast coffee
  Arms: Medium Roasted Coffee
Dietary Supplement: Dark Roasted Coffee — 12 oz dark roast coffee
  Arms: Dark Roasted Coffee

SUMMARY:
The present study determined the effects light, medium, and dark roasted, brewed coffees on blood glucose responses in normal (n = 19) subjects.

DETAILED DESCRIPTION:
This is a single-blinded, randomized partial block design conducted over 6 weeks in two parts.

In part 1 (3 weeks), participants were randomly assigned to consume four beverages: a placebo containing water and caramel color, light, medium, or dark roast coffee before, during, or after consumption of a beverage containing 50 g of glucose.

In part 2 (3 weeks), participants were randomly assigned to consume four beverages: a placebo containing water and caramel color, light, medium, or dark roast coffee before, during, or after consumption of a standardized breakfast (corn flakes cereal + skim milk) containing 50 g of glucose.

In each part, fasting and postprandial glucose profiles were determined.

ELIGIBILITY:
Inclusion Criteria:

• Age 18-64 years old with BMI less than 29 and fasting blood glucose less than 125 mg/dl.

Exclusion Criteria:

* Age 18-64 years old with BMI less than 29 and fasting blood glucose less than 125 mg/dl.
* Weight less than 110 pounds (55 kg)
* Pre-existing health conditions, such as:

  * High cholesterol
  * Hypertension
  * Cardiovascular disease
  * Gastrointestinal motility disorders
  * Hypo- or hyperthyroidism
  * Anemia
  * Renal disease
  * Liver disease, including hepatitis B or C, cholestasis, cirrhotic liver disease, or non-alcoholic fatty liver disease
  * Chronic or acute pancreatitis
  * Diabetes type 1 or 2
  * Insulin resistance
  * Polycystic ovary syndrome
* Food allergies or intolerances to coffee/caffeine/dairy/corn-based cereals.
* Currently taking prescription medication
* Current smoker
* Consumes more than 3 alcoholic beverages per day
* Pregnant or breastfeeding
* Not willing to take their own blood samples with finger sticks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Glucose | 6 weeks
  Each week, fasted baseline and postprandial measurements taken out to 240 minutes

SECONDARY OUTCOMES:
Changes in Glucose Area Under the Curve | 6 weeks
  Used glucose changes over 240 minutes to construct area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel K Harris, PhD, Principal Investigator — North Carolina State University
Locations (1):
- Schaub Hall, Campus Box 7624, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share IPD.

REFERENCES:
- [Derived] Rayo-Mendez LM, Kinzer C, McMahon J, Nguyen M, Harris GK. Coffee Roast Level, Timing, and Carbohydrate Source Affect Peak Blood Glucose and Area Under the Curve Values in a Randomized Pilot Clinical Trial. J Nutr Metab. 2025 Oct 23;2025:4174563. doi: 10.1155/jnme/4174563. eCollection 2025. PMID 41179392